CLINICAL TRIAL: NCT03260283
Title: Assessment of Subarachnoid Anesthesia With Low Dose of Pethidine and Combination of Ropivacaine With Fentanyl for Urologic Surgical Operations.
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Saint Savvas Anticancer Hospital (Other)
Responsible Party: Principal Investigator, Georgia Micha, Anesthesiologist,MD, MSc, PhD, Saint Savvas Anticancer Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: StSavvasAH 2
Record Dates: First submitted 2017-08-08; First posted 2017-08-24 (Actual); Last update posted 2020-03-31 (Actual); Status verified 2020-03

CONDITIONS: Low Dose of Pethidine for Subarachnoid Anesthesia
Keywords: pethidine
MeSH Terms: interventions — Meperidine; Fentanyl

STUDY DESIGN:
Intervention Model Description: Double blind randomized control trial
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (Experimental): 0.4 mgkg-1 of pethidine hydrochloride
  Interventions: Drug: Pethidine hydrochloride
- Group II (Experimental): 2ml of ropivacaine (0.75%) with 15 mcg of fentanyl
  Interventions: Drug: Ropivacaine HCl Inj 7.5 MG/ML; Drug: Fentanyl

INTERVENTIONS:
Drug: Pethidine hydrochloride — In Group I patients will be administered with low dose of pethidine hydrochloride (0.4 mgkg-1) diluted into normal saline up to 2 ml of total volume in order to perform subarachnoid anesthesia for urologic operations
  Arms: Group I
Drug: Ropivacaine HCl Inj 7.5 MG/ML — In Group II patients will be administered with 2 ml of ropivacaine (0.75%)
  Arms: Group II
Drug: Fentanyl — 15 mcg of fentanyl will be added to the solution in order to perform subarachnoid anesthesia for urologic operations
  Arms: Group II

SUMMARY:
The aim of this study is to assess the efficacy of subarachnoid anesthesia with low dose of pethidine (0.4mgkg-1) compared to administration of ropivacaine and fentanyl which is nowadays the common practice.

ELIGIBILITY:
Inclusion Criteria:

* All patients about to be subjected to Transurethral resection of the prostate (TURP) and Transurethral resection of urinary bladder tumors (TUR)
* Signed informed consent

Exclusion Criteria:

* When subarachnoid block is contraindicated
* Patient's denial in performing subarachnoid anesthesia
* Failure of subarachnoid block (L1 dermatome in 30 minutes after intrathecal drug administration)
* Mental illness or drug abuse
* Estimated time of operation >90 minutes

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2017-08-16 (Actual); Primary Completion 2018-11-29 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Efficacy of subarachnoid anesthesia after administration of low dose of pethidine hydrochloride as the sole anesthetic agent, assessed by the pinprick test. | 30 minutes after the intrathecal administration of the drug
  Low dose of pethidine hydrochloride will be administered for subarachnoid anesthesia in patients subjected to urologic operations.The level of sensory block after subarachnoid anesthesia will be assessed by the pinprick test.
Efficacy of subarachnoid anesthesia after administration of low dose of pethidine hydrochloride as the sole anesthetic agent, assessed by the modified Bromage scale. | 30 minutes after the intrathecal administration of the drug
  The level of motor block will be assessed by the modified Bromage scale.
Efficacy of subarachnoid anesthesia after administration of low dose of pethidine hydrochloride as the sole anesthetic agent, assessed by the time of motor block establisment. | 30 minutes after the intrathecal administration of the drug
  Time of motor block establishment (Grade 2 in modified Bromage scale) will be recorded as well as the time of withdrawal. Failure of spinal block is considered when there is no block at the level of first lumbar vertebra 30 minutes after the intrathecal administration of the drugs and in these cases the patients are excluded from the study.

SECONDARY OUTCOMES:
Efficacy and length of time of analgesia provided by the low dose of pethidine hydrochloride. | In the first 24 hours postoperatively
  In order to assess the efficacy of analgesia provided by the low dose of pethidine hydrochloride we record the time at which patients ask analgesic for the first time after the operation.
Percentage of postsurgical catheter-related bladder discomfort | Change from preoperative status to postoperative one at 0, 1, 2, 6, 24 hours postoperatively
  Assessment of discomfort will be made by a scale of four (1=no discomfort, 2=mild discomfort reported on questioning only, 3=moderate discomfort, urge to pass urine reported by the patient without questioning, 4= severe discomfort, urge to pass urine accompanied by behavioral responses, such as flailing limbs, strong vocal responses or attempts to pull the catheter out)
Assessment of haemodynamic status of patients intraoperatively | During the operation
  In order to assess the haemodynamic status of patients intraoperatively we record all episodes of hypotension (drop of systolic pressure >30% of value before the subarachnoid block.
Length of stay in postanesthesia care unit | Time of entry into postanesthesia care unit up to discharge to the ward or two hours time whichever comes first.
  We record the total amount of time that patients stay in the postanesthesia care unit immediately after the operation until they are discharged to the ward. In order for a patient to be discharged to the ward he must have a score of more than >9 in Aldrete's Scoring system.
Adverse events | All adverse events observed intraoperatively and in the first 24 hours postoperatively
  We record all adverse events observed intraoperatively and 24 hours postoperatively
Efficacy and length of time of analgesia provided by the low dose of pethidine hydrochloride. | In the first 24 hours postoperatively
  We also record the total amount of analgesics administered in morphine analogues in the first 24 hours postoperatively.
Assessment of haemodynamic status of patients intraoperatively | During the operation
  We also record the total amount of intravenous fluids administered intraoperatively.

CONTACTS AND LOCATIONS:
Overall Officials: Sofia Poulopoulou, Head of department, Study Director — Anticancer Hospital of Athens 'Saint Savvas'
Locations (1):
- Anticancer Hospital of Athens "Saint Savvas", Athens, Greece

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Luck JF, Fettes PD, Wildsmith JA. Spinal anaesthesia for elective surgery: a comparison of hyperbaric solutions of racemic bupivacaine, levobupivacaine, and ropivacaine. Br J Anaesth. 2008 Nov;101(5):705-10. doi: 10.1093/bja/aen250. Epub 2008 Sep 2. PMID 18765643
- [Background] Mohta M. Ropivacaine: Is it a good choice for spinal anesthesia? J Anaesthesiol Clin Pharmacol. 2015 Oct-Dec;31(4):457-8. doi: 10.4103/0970-9185.169050. No abstract available. PMID 26702199
- [Background] Lewis RP, Spiers SP, McLaren IM, Hunt PC, Smith HS. Pethidine as a spinal anaesthetic agent--a comparison with plain bupivacaine in patients undergoing transurethral resection of the prostate. Eur J Anaesthesiol. 1992 Mar;9(2):105-9. PMID 1555549